CLINICAL TRIAL: NCT03423407
Title: Evaluation of Attenuation Correction Accuracy in Positron Emission Tomography-Magnetic Resonance Imaging (PET-MRI)
Status: Terminated | Type: Observational
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201710134; 1R01CA212148-01 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: PET/CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PET/MR: * Participants will be scanned on a PET-MRI scanner which is FDA-approved and will operate within FDA-approved guidelines.
  * Participants will be asked to lie still within the scanner for up to 90 minutes
  Interventions: Device: Positron Emission Tomography-Magnetic Resonance Imaging (PET-MRI)

INTERVENTIONS:
Device: Positron Emission Tomography-Magnetic Resonance Imaging (PET-MRI) — FDA approved scanner
  Other Names: PET/MR; PET/MRI

SUMMARY:
The purpose of this research proposal is to establish a mechanism to develop tools that will allow the investigators to measure the impact of magnetic resonance (MR) acquisition correction sequences for attenuation correction on positron emission tomography (PET) quantitation accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age
* Participant can be a male or a non-pregnant female.
* Successful completion of MRI screening form
* Participant must have undergone a PET/CT examination with injection of a standard dose of 18F-fluorodeoxyglucose (FDG) or other PET tracer with a half-life greater than one hour either for clinical or research purposes within 3 hrs of the proposed PET-MRI examination.
* Participant will be fully informed and has personally signed and dated the written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) provisions

Exclusion Criteria:

* Subjects for whom exposure to a strong magnetic field would be a health risk (e.g., subjects with cardiac pacemakers or non-MR compatible metallic implants)
* Women who are pregnant.
* Subjects who require sedation to participate will be excluded.
* Patient/participant has a medical condition which in the judgment of the investigator might make supine positioning for the duration of the scan unsafe, such as (but not limited to) congestive heart failure or significant pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen at Washington University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Measure the impact of MR acquisition correction sequences for attenuation correction on PET quantitation accuracy | At the time of the MRI scan
  -PET images from PET/MRI with the MR derived attenuation correction will be compared to images generated with the CT attenuation correction from the standard of care PET/CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Laforest, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu